CLINICAL TRIAL: NCT05827393
Title: Muscle Transplantation for Large Angle Horizontal Strabismus: Esotropia Versus Exotropia
Brief Title: Muscle Transplantation in Strabismus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, doaa abody ahmed, assistant lecturer ophthalmology, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 155
Record Dates: First submitted 2023-02-19; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Strabismus, Noncomitant
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): 15 patients with large angle esotropia
  Interventions: Procedure: muscle transplantation
- group B (Active Comparator): 15 patients with large angle exotropia
  Interventions: Procedure: muscle transplantation

INTERVENTIONS:
Procedure: muscle transplantation — the resected extra stump of rectus muscle was transplanted to the other horizontal rectus muscle which was recessed by a standard recession technique

SUMMARY:
All the patients underwent standard muscle transplantation, where the resected extra stump of lateral or medial rectus muscle was transplanted to the medial or lateral rectus muscle using 6-0 prolene which wasrecessed by a standard recession technique

ELIGIBILITY:
Inclusion Criteria:

* Patients with esotropia or exotropia of more than 60 prism dioptre

Exclusion Criteria:

* Muscular paralysis.
* High myopia. .Dissociated vertical divergence. .Accommodative esotropias.
* Large vertical deviations associated Alphabetic syndromes
* previous surgeries in either eye

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-11 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Compare the angle of strabismus after muscle transplantation procedure in large angle esotropia with large angle exotropia | one day
  the change of angle of strabismus will be assessed pre and post muscle transplantation procedure , the angle of strabismus will be measured pre operative and postoperative after one day using hirschburg test measured by degree

SECONDARY OUTCOMES:
assess the angle of strabismus after muscle transplantation procedure in large angle esotropia with large angle exotropia | six months
  the stability of angle of strabismus will be assessed post muscle transplantation procedure , the angle of strabismus will be measured after six month post operative using hirschburg test measured by degree

CONTACTS AND LOCATIONS:
Locations (1):
- Qena University Hospital, Qina, Egypt